CLINICAL TRIAL: NCT02330133
Title: Mid-life Women: Preventing Unintended Pregnancy and STIs
Acronym: FemRepro_2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Lynne Swartz, Research Scientist, Oregon Center for Applied Science, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SBIR64R-2; R44HD044374 (NIH)
Record Dates: First submitted 2010-05-04; First posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Reproductive Health
Keywords: mid-life women; unintended pregnancy; STI/HIV prevention; intervention; interactive; CD-ROM; multimedia; video

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Women's Reproductive Health (Experimental): Targeted text and video information on website for women aged 25-55 to avoid unplanned pregnancy and sexually transmitted infections
  Interventions: Behavioral: Women's Reproductive Health
- Online sexual health content (Active Comparator): Online general text-based information about reproductive health issues and STD prevention strategies
  Interventions: Behavioral: Online sexual health content

INTERVENTIONS:
Behavioral: Women's Reproductive Health — Targeted text and video information on website for women aged 25-55 to avoid unplanned pregnancy and sexually transmitted infections
  Other Names: Women's Reproductive Health: A Guide to Staying Healthy
  Arms: Women's Reproductive Health
Behavioral: Online sexual health content — Online general text-based information about reproductive health issues and strategies for preventing sexually transmitted infections
  Arms: Online sexual health content

SUMMARY:
Mid-life women, aged 35-50, are currently an underserved population in the areas of unintended pregnancy and STI prevention interventions. Common perception is that women in this age range are no longer sexually active, or are past the menopause transition, but in reality, sexual activity remains stable through mid-life and into the post-menopausal years. Additionally, physiological and relationship status changes (e.g. divorce or death of a partner) put these women at increased risk for both unintended pregnancy and STI's. This project developed and evaluated a theoretically-based multimedia intervention designed to assist mid-life women in protecting themselves from sexually transmitted infections and unintended pregnancy.

DETAILED DESCRIPTION:
The primary aim of this project was to create and evaluate a theoretically-based, interactive multimedia program for women aged 35-55 to assist them in avoiding unintended pregnancy and sexually transmitted infections (STIs). The intervention, titled "Women's Reproductive Health: A guide to staying healthy," addressed these concerns across the life span and was designed to increase knowledge about (a) pregnancy risk; (b) STI risk; (c) strategies to prevent STIs and unintended pregnancy; (d) influences of sexual partners on risk reduction decisions and behaviors; (e) partner communication techniques; and (f) health care provider communication techniques.Overall features of the program include video, interactive tools, animations, text information pages, and various links both across and within specific modules to link related information. A feature titled "My Notes" allowed the user to save content from the program into an easily retrievable repository.

Motivational videos featuring friendly mid-life hosts could be viewed on the first page of each module, as well as on the home page and topic introduction pages. These videos not only provided specific information about the content, they also provided message framing and set the tone of the program segment. Other videos included testimonials on topics such as contraceptive methods, sexually transmitted infections, and other health information. Interactive materials include an assessment checklist for STI risk, a quiz to help the user identify the types of birth control methods that best fit her lifestyle and preferences, as well as several checklists

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25-55.

Exclusion Criteria:

* Males
* Women under 25 years of age and over 55

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 333 (Actual)
Dates: Start 2008-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Knowledge of reproductive health issues | 7-day posttest and 30-day follow-up
  A 22-item knowledge scale was created to assess content areas of the program (e.g., 3 items on anatomy & physiology, 16 items on pregnancy prevention, and 4 items on STI prevention). For example, users were asked to answer the question "A women is most likely to become pregnant (no matter how long or short her menstrual cycle) if she has sexual intercourse about:" with choices being (a) 1 week before menstruation beings, (b) 2 weeks after menstruation begins, (c) 2 weeks before menstruation begins, (d) 1 week after menstruation begins, or (e) do not know.

SECONDARY OUTCOMES:
Attitudes about reproductive health and prevention | 7-day posttest and 30-day follow-up
  Participant attitudes were measured using scales that assessed the perceived importance of using a contraceptive method to prevent pregnancy (6 items), the perceived importance of talking with your partner about contraception (4 items) and two additional items measuring the perceived importance of using a contraceptive method to prevent STIs (1 item), and the perceived importance of talking with your healthcare provider (1 item) (alpha =.74, test- retest reliability=.73).
Self-efficacy for engaging in strategies to prevent pregnancy and communicate with partner about health risks | 7-day posttest and 30-day follow-up
  Participant self-efficacy was measured using scales that assessed confidence in preventing pregnancy (6 items), and talking with the partner (2 items) (alpha=84, test-retest reliability=.68).
Intentions to engage in strategies to prevent pregnancy and communicate with | 7-day posttest and 30-day follow-up
  Participant behavioral intentions were measured using scales that assessed intention of using a contraceptive method (2 items), preventing an STI (4 items), and talking with a sexual partner (4 items) (alpha=.74, test-retest reliability=.69).

CONTACTS AND LOCATIONS:
Overall Officials: Lynne H Grilley Swartz, MPH, CHES, Principal Investigator — Oregon Center for Applied Science
Locations (1):
- Oregon Center for Applied Science, Eugene, Oregon, United States